CLINICAL TRIAL: NCT01744665
Title: A Phase II Randomized, Multicenter Study of Treatment-free Remission in Chronic Myeloid Leukemia in Chronic Phase (CML-CP) Patients Who Achieve and Sustain MR4.5 After Switching to Nilotinib
Brief Title: A Study That Switched Patients From Imatinib to Nilotinib and Then Was Followed by Treatment Cessation
Acronym: ENESTgoal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AUS37
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: CML
Keywords: CML, chronic myeloid leukemia, stop, niotinib, discontinue, imatinib, switch, MR4.5, undetectable, bcr-abl
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Free Remission (Experimental): Patients entered a monitoring phase for 2 years and received 300 mg nilotinib mg bid. Patients who achieved MR4.5 entered a Consolidation Phase and were treated with nilotinib for 2 years. If MR4.5 was sustained during the Consolidation phase, patients were eligible to stop taking niltoinib during the treatment-free remission (TFR) phase.
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — Nilotinib will be provided as 150 mg capsules. Patients will take nilotinib 300mg twice daily on study and dose modifications to 450mg once daily is permitted per protocol.
  Other Names: AMN107

SUMMARY:
To evaluate molecular relapse free rates 6 months after stopping nilotinib therapy in patients who achieve MR4.5

DETAILED DESCRIPTION:
Study protocol included criteria for study termination that was met when > 2 patients lost CCyR during TFR phase (> 1% BCR-ABL); This study was terminated early as > 2 cases of confirmed loss of complete cytogenetic response were reported despite BCR-ABL monitoring during the TFR Phase. All cases achieved MR4.5 after Nilotinib treatment re-initiation and maintained until end of study; trial did not mandate re-initiation within 4 weeks after loss of MMR_ that was a requirement in other Nilotinib TFR trials Initial sample size was 300 patients with CML-CP; Amendment #2 in June 2015 reduced sample size to 59 due to recruitment challenges; Study endpoint analysis and interpretations of data were challenging due to small sample size for early study closure..

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CML
* Treated with at least 1 year of imatinib
* Bcr-Abl level by PCR must be less than or equal to 0.1% and greater than 0.0032% by PCR reported on the International scale confirmed during screening
* Written informed consent obtained prior to any screening procedures performed

Exclusion Criteria:

* T315I mutation
* Prior imatinib failure or had accelerated phase or blast crisis CML
* Impaired cardiac function
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-08-12 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (54):
- United States (54):
  - University of Alabama Comprehensive Cancer Center University of Alabama (8), Birmingham, Alabama
  - Banner MD Anderson Cancer Center Banner MD Anderson (2), Gilbert, Arizona
  - Scottsdale Healthcare/TGen Clinical Research Service SC, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - City of Hope National Medical Center Dept of Oncology, Duarte, California
  - Compassionate Care Research Group Inc CCCMG, Fountain Valley, California
  - UC San Diego UC San Diego Cancer Ctr, La Jolla, California
  - Wilshire Oncology Medical Group Corona Cancer Center, Multiple Locations, California
  - Epic-Care, Pleasant Hill, California
  - Sutter Institute for Medical Research Oncology/Hematology, Sacramento, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Rocky Mountain Cancer Centers USOR, Boulder, Colorado
  - Florida Cancer Specialists DeptofFloridaCancerSpecialists, Fort Myers, Florida
  - MD Anderson Cancer Center - Orlando Cancer Center, Orlando, Florida
  - H Lee Moffitt Cancer Center and Research Institute H. Lee Moffitt Cancer Ctr (67), Tampa, Florida
  - Stroger Cook County Hospital Division of Hematology & Onc, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics Holden Comprehensive Cancer Ct, Iowa City, Iowa
  - University of Kansas Hospital and Medical Center Clinical Research Center, Kansas City, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Christus Schumpert Health System, Shreveport, Louisiana
  - Michigan State University / Breslin Cancer Center Breslin Cancer Center (3), Lansing, Michigan
  - Billings Clinic Billings Clinic (8), Billings Montana, Montana
  - Hackensack University Medical Center John Theurer Cancer Center, Hackensack, New Jersey
  - Hematology Oncology Associates of Northern New Jersey PA Dept of Hem-Onc of Northern NJ, Morristown, New Jersey
  - Memorial Sloan Kettering Memorial Sloan Kettering (63), New York, New York
  - Weill Cornell Medical Center Dept. of Oncology, New York, New York
  - Columbia University Medical Center Herbert Irving Pavilion, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center Montefiore Medicial Center, The Bronx, New York
  - Westchester Medical Center NY Medical College, Valhalla, New York
  - Duke University Medical Center Duke University Med Ctr, Durham, North Carolina
  - Carolina Oncology Specialists, PC, Hickory, North Carolina
  - Wake Forest University Health Sciences Hematology and Oncology, Winston-Salem, North Carolina
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital OSU Medical Center, Columbus, Ohio
  - Northwest Cancer Specialists Compass Oncology -BKM, Portland, Oregon
  - University of South Carolina-Hollings Cancer Center Medical University of SC, Columbia, South Carolina
  - Tennessee Oncology Dept. of Centennial Medical, Nashville, Tennessee
  - Vanderbilt Univeristy Ingram Cancer Center (10), Nashville, Tennessee
  - Hendrick Cancer Center Hendricks Cancer Center, Abilene, Texas
  - Texas Oncology Texas Oncology - McAllen, Dallas, Texas
  - Texas Oncology Texas Oncology - Plano West, Dallas, Texas
  - Texas Oncology P A Texas Oncology - Midland, Dallas, Texas
  - University of Texas Medical Branch SC, Galveston, Texas
  - Oncology Consultants Oncology Consultants, P.A., Houston, Texas
  - The Methodist Hospital Cornell University, Houston, Texas
  - South Texas Cancer Center- McAllen, McAllen, Texas
  - Brooke Army Medical Center Brooke Army Medical, San Antonio, Texas
  - Waco Cancer and Research Center, Waco, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman Cancer Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Kadlec Clinic Hematology and Oncology SC, Kennewick, Washington
  - West Virginia University/ Mary Babb Randolph Cancer Center Mary Babb Randolph Cancer Ctr, Morgantown, West Virginia
  - Medical College of Wisconsin Med College of WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nilotinib: All patients enrolled in trial
Period: Monitoring Phase
Arm/Group | Nilotinib
Started | 59
Completed | 41
Not Completed | 18
Not completed — Adverse Event | 4
Not completed — Abnormal laboratory value(s) | 1
Not completed — Unsatisfactory therapeutic effect | 7
Not completed — Withdrawal by Subject | 5
Not completed — Did not achieve MR4.5 | 1
Period: Consolidation Phase
Arm/Group | Nilotinib
Started | 41
Completed | 22
Not Completed | 19
Not completed — Adverse Event | 2
Not completed — Unsatisfactory therapeutic effect | 4
Not completed — Withdrawal by Subject | 4
Not completed — Administrative problems | 9
Period: Treatment Free Remission Phase
Arm/Group | Nilotinib
Started | 32
Completed | 32
Not Completed | 0
Period: Re-initiation Phase
Arm/Group | Nilotinib
Started | 17
Completed | 4
Not Completed | 13
Not completed — Administrative problems | 10
Not completed — Adverse Event | 1
Not completed — No longer required treatment | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall: Patients entered a monitoring phase for 2 years and received 300 mg nilotinib mg bid. Patients who achieved MR4.5 entered a Consolidation Phase and were treated with nilotinib for 2 years. If MR4.5 was sustained during the Consolidation phase, patients were eligible to stop taking niltoinib during the treatment-free remission (TFR) phase.
Arm/Group | Overall
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 25
  Black | 2
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Molecular Relapse Within 6 Months After Starting the TFR Phase
Description: Percentage of particpants without confirmed loss of MMR within 6 months following nilotinib TFR is calculated by dividing the number of patients with no documented confirmed loss of MR4, in the first 6 months after starting nilotinib TFR phase by the number of patients who entered nilotinib TFR phase. Molecular relapse is defined as having a confirmed BCR-ABL ratio above MMR (2 consecutive BCR-ABL levels >0.1% IS taken approximately 4 weeks apart).
Time Frame: 6 months after stopping nilotinib therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 32
Participants
  Number of participants | 12

2. Secondary Outcome: Relapse Free Survival is Defined as Time From the Date of Nilotinib Treatment Discontinuation to the First Documented Molecular Relapse (Confirmed Loss of MR4.5).
Description: Relapse-free survival after the start of the TFR phase was summarized using the product-limit (Kaplan-Meier) estimates. The median for the relapse free survival and its 95% confidence intervals were provided. This analysis was performed on the FAS. Patients who dropped out without relapse were treated as censored observations.
Time Frame: 7 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 32
weeks | 21.4 [17.1 to NA] — The upper limit CI was not estimable

3. Secondary Outcome: Percentage of Participants Without Molecular Relapse Within 12 and 24 Months After Starting the Treatment -Free Remission (TFR) Phase
Description: The percentage of participants without confirmed loss of MRR at 12 and 24 months is calculated by dividing the number of patients with no documented confirmed loss of MR4 at 12 and 24 months after starting the nilotinib TFR phase by the number of patients who entered nilotinib TFR phase.
Time Frame: 12 and 24 months after starting the TFR
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 32
Participants
  Month 12: Number of participants | 8
  Month 24: Number of participants | 2

4. Secondary Outcome: Percentage of Participants Who Regained MR4.5 After Restarting Nilotinib Due to Molecular Relapse
Description: The percentage of participants who regained MR4.5 after restarting nilotinib will be calculated as the number of patients who achieved MR4.5 after having lost MR4 divided by the number of patients who lost MR4.
Time Frame: Restart of nilotinib up to month 6, 12 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 17
Participants
  Month 6: Number of participants | 7
  Month 12: Number of participants | 17
  Month 24: Number of participants | 17

5. Secondary Outcome: Number of Participants Who Progressed to Accelerated Phase/Blastic Crisis (AP/BC) or Died From From Any Cause.
Description: Progression to AP/BC and death where the "failure" event is the earliest occurrence of the following event: progression to AP/BC date.
Time Frame: Baseline up to approximately 5 years
Measure: Number; unit: participants
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 32
participants | 0

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of cessation of nilotinib therapy to the date of death from any cause.
Time Frame: Baseline up to approximately 5 years
Measure: Number; unit: participants
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 32
participants | 0

7. Secondary Outcome: Change in Symptom-burden Scores by the M.D. Anderson Symptom Inventory - Chronic Myeloid Leukemia (MDASI-CML) Assessment
Description: The M.D. Anderson Symptom Inventory for CML patients (MDASI-CML) was used to assess the nature and impact of symptom burden on life. It consisted of 20 validated symptom items and 6 validated interference items. Each item was assessed on an 11 point scale with responses from 0-10, 0=not present and 10=as bad as you can imagine. Symptom score (SS) was calculated when a patient scored at least 8 items of the symptom items using the formula: (sum of scores for the items answered) / number of items answered. If a subject responded to < 8 symptom items, the score was considered missing. Interference score (IS) was calculated when a patient scored at least 4 items using the formula: (sum of scores for the items answered)/number of items answered. If a subject responded to < 4 interference items, the score was considered missing. The total symptom score was 0-200 and total interference score was 0-60. Mean change from baseline was summarized at all post-baseline time points
Time Frame: From baseline to time to when MR4.5 is confirmed, up to 24 months, and from end of Consolidation Phase to 6 and 12 months into the TFR Phase
Population: Number of participants who completed questionnaire varied across visits
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 59
scores on a scale
  SS Baseline (observed value), n=40: number analyzed (Participants) | 40
  SS Baseline (observed value), n=40 | 0.125 (0.1314)
  SS Consolidation Ph - M 3 (change from BL) n=26: number analyzed (Participants) | 26
  SS Consolidation Ph - M 3 (change from BL) n=26 | 0.012 (0.1362)
  SS Consolidation Ph - M 12 (change from BL) n=30: number analyzed (Participants) | 30
  SS Consolidation Ph - M 12 (change from BL) n=30 | 0.021 (0.1140)
  SS Consolidation Ph - M 24 (change from BL) n=26: number analyzed (Participants) | 26
  SS Consolidation Ph - M 24 (change from BL) n=26 | 0.026 (0.1402)
  SS TFR Baseline (observed value) n=32: number analyzed (Participants) | 32
  SS TFR Baseline (observed value) n=32 | 0.160 (0.1496)
  SS TFR - Month 6 (change from BL) n=10: number analyzed (Participants) | 10
  SS TFR - Month 6 (change from BL) n=10 | -0.005 (0.1773)
  SS TFR - Month 12 (change from BL) n=5: number analyzed (Participants) | 5
  SS TFR - Month 12 (change from BL) n=5 | -0.032 (0.1034)
  IS Baseline (observed value), n=40: number analyzed (Participants) | 40
  IS Baseline (observed value), n=40 | 0.123 (0.2156)
  IS Consolidation Ph - M 3 (change from BL) n=25: number analyzed (Participants) | 25
  IS Consolidation Ph - M 3 (change from BL) n=25 | 0.008 (0.1911)
  IS Consolidation Ph - M 12 (change from BL) n=30: number analyzed (Participants) | 30
  IS Consolidation Ph - M 12 (change from BL) n=30 | -0.005 (0.1983)
  IS Consolidation Ph - M 24 (change from BL) n=26: number analyzed (Participants) | 26
  IS Consolidation Ph - M 24 (change from BL) n=26 | 0.015 (0.1942)
  IS TFR Baseline (observed value) n=32: number analyzed (Participants) | 32
  IS TFR Baseline (observed value) n=32 | 0.141 (0.2067)
  IS TFR - Month 6 (change from BL) n=10: number analyzed (Participants) | 10
  IS TFR - Month 6 (change from BL) n=10 | -0.015 (0.1780)
  IS TFR - Month 12 (change from BL) n=5: number analyzed (Participants) | 5
  IS TFR - Month 12 (change from BL) n=5 | -0.037 (0.1880)

8. Secondary Outcome: Change in Health Utility Assessed by EuroQol Group-5D-3L (EQ-5D-3L) Visual Analogue - Safety Set
Description: The EQ-5D-3L questionnaire comprises 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and visual analog has a scale 0 to 100 (0=worst imaginable health state, 100=best imaginable health state).
Time Frame: From baseline to time to when MR4.5, up to 24 months, is confirmed and from end of Consolidation Phase to 6 and 12 months into the TFR Phase
Population: Number of participants who completed questionnaire varied across visits
Measure: Median (Full Range); unit: scores on scale
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 36
scores on scale
  Baseline (observed value) | 83.250 [4.50 to 100.00]
  Consolidation Ph - M 3 (change from BL): number analyzed (Participants) | 24
  Consolidation Ph - M 3 (change from BL) | 2.000 [-50.00 to 87.00]
  Consolidation Ph - M 12 (change from BL): number analyzed (Participants) | 31
  Consolidation Ph - M 12 (change from BL) | 3.250 [-75.00 to 82.00]
  Consolidation Ph - M 24 (change from BL): number analyzed (Participants) | 28
  Consolidation Ph - M 24 (change from BL) | 1.350 [-30.00 to 85.50]
  TFR Baseline (observed value): number analyzed (Participants) | 32
  TFR Baseline (observed value) | 80.00 [9.35 to 100.00]
  TFR - Month 6 (change from BL): number analyzed (Participants) | 9
  TFR - Month 6 (change from BL) | 10.00 [-30.00 to 89.65]
  TFR - Month 12 (change from BL): number analyzed (Participants) | 5
  TFR - Month 12 (change from BL) | 0.000 [-20.00 to 35.00]

9. Secondary Outcome: Change in Observed Scores for Patient Quality of Life Assessed by SF-8 - Safety Set
Description: The SF-8 questionnaire consisted of 8 items (general health, physical functioning, role physical, bodily pain, vitality, social functioning, role-emotional and mental health) and was used to assess the impact of nilotinib treatment discontinuation on the quality of life. Each item had a 1 to 5 or 1 to 6 point response range and the higher number in the raw scores indicated poorer quality of life. The physical and mental component summary measures were calculated using a norm-based scoring method given in the instrument guidelines. These norm-based scores were summarized at baseline and mean change from baseline for post-baseline time points. The norm-based scores (based on the US population) had a mean of 50 and standard deviation of 10. Higher norm-based summary scores indicated better health
Time Frame: From baseline to time to when MR4.5 is confirmed and from end of Consolidation Phase to 6 and 12 months into the TFR Phase
Population: Number of participants who completed questionnaire varied across visits
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Free Remission
Number analyzed (Participants) | 41
scores on a scale
  Baseline | 50.508 (8.4313)
  Consolidation Ph - M 3: number analyzed (Participants) | 26
  Consolidation Ph - M 3 | 50.720 (7.6047)
  Consolidation Ph - M 12: number analyzed (Participants) | 31
  Consolidation Ph - M 12 | 49.020 (10.1851)
  Consolidation Ph - M 24: number analyzed (Participants) | 28
  Consolidation Ph - M 24 | 47.648 (8.7416)
  TFR Baseline: number analyzed (Participants) | 32
  TFR Baseline | 48.382 (8.6503)
  TFR - Month 6: number analyzed (Participants) | 9
  TFR - Month 6 | 46.605 (9.5042)
  TFR - Month 12: number analyzed (Participants) | 5
  TFR - Month 12 | 46.006 (8.6997)

10. Secondary Outcome: Percentage of Participants' Scores at Each Level Assessed by EQ-5D-3L for Month 3 in Consolidation Phase - Safety Set
Description: The EuroQol Five Dimensional Three-level (EQ-5D-3L) questionnaire comprises 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each item has 3 levels (no problems, some problems and extreme problems). The percentages of patients at each level of the five items of the EQ-5D-3L will be summarized at each time point
Time Frame: At month 3 in Consolidation Phase
Population: all completers did not complete all categories of questionaire
Measure: Count of Participants; unit: Participants
Groups:
- No Problems: No problems
- Some Problems: Some problems
- Extreme Problems: Extreme problems
Arm/Group | No Problems | Some Problems | Extreme Problems
Number analyzed (Participants) | 26 | 26 | 26
Participants
  Mobility: Number of participants | 22 | 4 | 0
  Self-Care: Number of participants | 25 | 1 | 0
  Usual Activities: Number of participants | 21 | 5 | 0
  Pain/Discomfort: number analyzed (Participants) | 25 | 25 | 25
  Pain/Discomfort: Number of participants | 12 | 13 | 0
  Anxiety / Depresssion: Number of participants | 20 | 6 | 0

11. Secondary Outcome: Percentage of Participants' Scores at Each Level Assessed by EQ-5D-3L for Month 12 in Consolidation Phase - Safety Set
Description: as for outcome 10
Time Frame: Month 12 in Consolidation Phase
Population: all completers did not complete all categories of questionaire
Measure: Count of Participants; unit: Participants
Arm/Group | No Problems | Some Problems | Extreme Problems
Number analyzed (Participants) | 31 | 31 | 31
Participants
  Mobility: Number of participants | 23 | 8 | 0
  Self-Care: Number of participants | 31 | 0 | 0
  Usual Activities: Number of participants | 23 | 7 | 1
  Pain/Discomfort: number analyzed (Participants) | 30 | 30 | 30
  Pain/Discomfort: Number of participants | 18 | 11 | 1
  Anxiety / Depresssion: Number of participants | 21 | 10 | 0

12. Secondary Outcome: Percentage of Participants' Scores at Each Level Assessed by EQ-5D-3L for Month 24 in Consolidation Phase - Safety Set
Description: as for outcome 10
Time Frame: Month 24 in Consolidation Phase
Population: all completers did not complete all categories of questionaire
Measure: Count of Participants; unit: Participants
Arm/Group | No Problems | Some Problems | Extreme Problems
Number analyzed (Participants) | 28 | 28 | 28
Participants
  Mobility: number analyzed (Participants) | 27 | 27 | 27
  Mobility: Number of participants | 19 | 8 | 0
  Self-Care: Number of participants | 28 | 0 | 0
  Usual Activities: number analyzed (Participants) | 27 | 27 | 27
  Usual Activities: Number of participants | 23 | 4 | 0
  Pain/Discomfort: Number of participants | 17 | 9 | 2
  Anxiety / Depresssion: number analyzed (Participants) | 27 | 27 | 27
  Anxiety / Depresssion: Number of participants | 19 | 8 | 0

13. Secondary Outcome: Percentage of Participants' Scores at Each Level Assessed by EQ-5D-3L for Month 6 in Treatment Free Remission Phase - Safety Set
Description: The EuroQol Five Dimensional Three-level questionnaire (EQ-5D-3L) comprises 5 items: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each item has 3 levels (no problems, some problems and extreme problems). The percentages of patients at each level of the five items of the EQ-5D-3L will be summarized at each time point
Time Frame: Month 6 in in Treatment Free Remission Phase
Population: all completers did not complete all categories of questionaire
Measure: Count of Participants; unit: Participants
Arm/Group | No Problems | Some Problems | Extreme Problems
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Mobility: Number of participants | 7 | 3 | 0
  Self-Care: Number of participants | 10 | 0 | 0
  Usual Activities: Number of participants | 10 | 0 | 0
  Pain/Discomfort: Number of participants | 5 | 4 | 1
  Anxiety / Depresssion: Number of participants | 8 | 2 | 0

14. Secondary Outcome: Percentage of Participants' Scores at Each Level Assessed by EQ-5D-3L for Month 12 in Treatment Free Remission Phase - Safety Set
Description: as for outcome 13
Time Frame: Month 12 in in Treatment Free Remission Phase
Population: all completers did not complete all categories of questionaire
Measure: Count of Participants; unit: Participants
Arm/Group | No Problems | Some Problems | Extreme Problems
Number analyzed (Participants) | 5 | 5 | 5
Participants
  Mobility: Number of participants | 4 | 1 | 0
  Self-Care: Number of participants | 5 | 0 | 0
  Usual Activities: Number of participants | 4 | 1 | 0
  Pain/Discomfort: Number of participants | 1 | 4 | 0
  Anxiety / Depresssion: Number of participants | 3 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment or last day in TFR Phase up to approximately 5 years
Groups:
- Nilotinib: Nilotinib
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 19/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=59)
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Device embolisation (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Vascular stent stenosis (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Vascular headache (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Leg amputation (Surgical and medical procedures) | 1
Arterial stenosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=59)
Palpitations (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 3
Dry eye (Eye disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 23
Influenza like illness (General disorders) | 4
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 3
Pyrexia (General disorders) | 4
Bronchitis (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 5
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 4
Blood cholesterol increased (Investigations) | 5
Lipase increased (Investigations) | 11
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT01744665/SAP_000.pdf
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT01744665/Prot_001.pdf